CLINICAL TRIAL: NCT00442676
Title: Clinical Trial of a COX-2 Inhibitor for the Treatment of Women With Preeclampsia
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: No patients were recruited. Treatment drug expired.
Sponsor: Virginia Commonwealth University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: VCU IRB HM10590
Record Dates: First submitted 2007-02-28; First posted 2007-03-02 (Estimated); Last update posted 2012-03-13 (Estimated); Status verified 2012-03

CONDITIONS: Preeclampsia
MeSH Terms: conditions — Pre-Eclampsia | interventions — Celecoxib

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): Celecoxib, 200 mg/day
  Interventions: Drug: Celecoxib
- 2 (Placebo Comparator): Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Celecoxib — Capsule, 200 mg/day until 32 weeks of gestation
  Other Names: Celebrex
  Arms: 1
Drug: Placebo — Gelatin capsules of lactose
  Arms: 2

SUMMARY:
Preeclampsia is a hypertensive disorder of pregnancy and a leading cause of fetal and maternal morbidity and mortality. Recent findings indicate preeclampsia is an inflammatory disorder associated with increased expression of COX-2. This study will test the hypothesis that treatment of women with a COX-2 inhibitor, celecoxib, will stop the inflammatory process and reverse symptoms of preeclampsia.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women with preeclampsia between 20 - 32 weeks gestation. Preeclampsia is defined as a maternal blood pressure of >140/90 mmHg on two readings at least 6 hours apart with proteinuria of >300 mg/24 hours.

Exclusion Criteria:

* Exclusion criteria includes patients with known sensitivity to celecoxib; patients who have demonstrated allergic-type reactions to sulfonamides; patients who have experienced asthma, urticaria, or allergic-type reactions after taking aspirin or other NSAIDs. Other exclusion criteria will include patients with known cardiovascular disease or risk factors for cardiovascular disease, a prior history of ulcer disease or GI bleeding, impaired renal function, or liver dysfunction. Exclusion criteria will also include concomitant use of oral corticosteroids, anticoagulants, diuretics, ACE inhibitors, aspirin, fluconazole, and lithium.

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2009-06; Primary Completion 2010-01 (Actual); Study Completion 2010-01 (Actual)

PRIMARY OUTCOMES:
Length from start of treatment to delivery | From start of treatment to delivery

SECONDARY OUTCOMES:
Prevalence of severe preeclampsia | From start of treatment to delivery
Blood pressure | From start of treatment to delivery
Proteinuria | From start of treatment to delivery
Maternal complications | From start of treatment to delivery
Fetal/neonatal status | From start of treatment to delivery
Gestational age at delivery | At time of delivery
Birth weight | At time of delivery

CONTACTS AND LOCATIONS:
Overall Officials: Scott W Walsh, PhD, Principal Investigator — Virginia Commonwealth University; Susan M Lanni, MD, Study Director — Virginia Commonwealth University; Fidelma B Rigby, MD, Study Director — Virginia Commonwealth University; Nicole W Karjane, MD, Study Director — Virginia Commonwealth University
Locations (1):
- MCV Main Hospital, Richmond, Virginia, United States

REFERENCES:
- [Background] Shah TJ, Walsh SW. Activation of NF-kappaB and expression of COX-2 in association with neutrophil infiltration in systemic vascular tissue of women with preeclampsia. Am J Obstet Gynecol. 2007 Jan;196(1):48.e1-8. doi: 10.1016/j.ajog.2006.08.038. PMID 17240230
- [Background] Leik CE, Walsh SW. Neutrophils infiltrate resistance-sized vessels of subcutaneous fat in women with preeclampsia. Hypertension. 2004 Jul;44(1):72-7. doi: 10.1161/01.HYP.0000130483.83154.37. Epub 2004 May 17. PMID 15148293
- [Background] Groom KM, Shennan AH, Jones BA, Seed P, Bennett PR. TOCOX--a randomised, double-blind, placebo-controlled trial of rofecoxib (a COX-2-specific prostaglandin inhibitor) for the prevention of preterm delivery in women at high risk. BJOG. 2005 Jun;112(6):725-30. doi: 10.1111/j.1471-0528.2005.00539.x. PMID 15924527